CLINICAL TRIAL: NCT06904001
Title: Study on the Construction and Application of Early Warning Model of Sepsis in Critically Ill Patients
Acronym: sepsis model
Status: Enrolling by invitation | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHOWMU-CR2018-11-129
Record Dates: First submitted 2025-03-11; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Sepsis; Sepsis and Septic Shock; Infection
Keywords: sepsis; septic shock; biomarker; warning model
MeSH Terms: conditions — Sepsis; Shock, Septic; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — When admitted to the ICU, 1 ml of whole blood was collected, leukocyte mRNA was extracted, reverse transcribed, and stored in a -80℃ specimen bank.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sepsis and control: The presence of sepsis at the time of admission to the ICU is called sepsis, and the absence of sepsis is called control.

SUMMARY:
The condition of sepsis patients changes rapidly, whom are often accompanied by impaired respiratory, circulatory, renal, and coagulation functions. So far, the prognosis of sepsis at home and abroad is not ideal. Participants was randomly included in this research project on the pathogenesis and prevention of sepsis due to typical sepsis symptoms. the investigators will collect appropriate clinical specimens for analysis of immune cell functions and pathogenic microorganisms combined with individual patient research. This study will enable sepsis patients to be identified early and receive earlier anti-sepsis treatment, which is expected to improve the prognosis of sepsis, shorten hospitalization time, and reduce treatment costs.

The above-mentioned tests and analyses do not increase the economic burden on the participants, and the required expenses are all paid from the project funds; they do not affect the prognosis and rehabilitation process of participants, and do not have adverse effects on the health of participants.

ELIGIBILITY:
Inclusion Criteria:

1. Temperature > 38°C or < 36°C;
2. Heart rate > 90 beats/min;
3. Respiratory rate > 20 breaths/min or PaCO₂ < 32 mmHg;
4. White blood cell count > 12.0 × 10⁹/L or < 4.0 × 10⁹/L, or > 10% immature neutrophils;
5. Initial septic shock diagnosis;
6. Organ dysfunction (cardiovascular, respiratory, or ≥ 2 other organs);
7. Complete clinical data.

Exclusion Criteria:

1. Cancer history;
2. Chemotherapy;
3. Radiotherapy;
4. Incomplete data.
5. Controls were free of infectious or inflammatory diseases and glucocorticoid use.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU with sepsis, aged over 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Death | From the date of first ICU admission to the date of ICU discharge (whether due to death or clinical improvement), assessed up to 90 days.
  Whether death occurred during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Protecting patient privacy